CLINICAL TRIAL: NCT00858026
Title: Impact of a Fermented Infant Formula in Weaning Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bledina (Industry)
Collaborators: MAPI (Unknown)
Responsible Party: Valérie Brenas, Bledina
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: BL009
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Weaning
Keywords: weaning; breastfeeding; infant formula; fermented formula
MeSH Terms: conditions — Breast Feeding | interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Breastfed babies
  Interventions: Other: Breastmilk
- 2 (Active Comparator): Weaning with the standard milk
  Interventions: Other: Standard milk
- 3 (Experimental): Weaning with the fermented milk
  Interventions: Other: Fermented milk

INTERVENTIONS:
Other: Breastmilk — Exclusively breastfed babies
  Other Names: No other names
  Arms: 1
Other: Standard milk — Weaning babies fed with the standard formula
  Other Names: No other names
  Arms: 2
Other: Fermented milk — Weaning babies fed with the fermented formula
  Other Names: No other names
  Arms: 3

SUMMARY:
When mothers wanted to shift from breast milk to infant formulae, babies were randomly assigned to receive a fermented or a standard formula. Biological and clinical investigations were achieved at baseline (V1), and after one (V2) and three months (V3) of consumption of study formula. Intestinal microbiota was assessed by using culture-dependent techniques.

ELIGIBILITY:
Inclusion Criteria:

* Eutrophic infants, (± 2SD), healthy, male or female, of 2 months of age (± 1 week)
* Born at 37 weeks of amenorrhea or more
* Exclusively breastfed since birth
* Written informed consent given by both parents (or tutors) for study participation
* Parents (or tutors) agreeing on the follow-up by one of the study investigators

Exclusion Criteria:

* Infant with congenital or acquired immunodeficiency, whatever the aetiology
* Infant with a significant metabolic, organic or bowel disease which could interfere with the results of the present study,
* Infant with congenital and/or chromosomal malformation,
* Infant having received antibiotic therapy within the 3 weeks before the inclusion visit
* infant receiving a treatment susceptible to interfere with the measure of study parameters
* Antibiotic therapy per/pre/post partum > 48 h
* Infant needing the prescription of a specific milk (HA, without cow milk)
* Infant in a situation which could interfere with an optimal participation to the study, or which could represent a risk for the infant, according to the investigator.

Ages: 54 Days to 68 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine the impact of a fermented infant formula on the intestinal microbiota in weaning babies | 2, 3 and 5 months of age

SECONDARY OUTCOMES:
Describe the intestinal flora according to the nutrition group | 3 and 5 months of age
Compare the effect on enterobacteria and clostridium of a fermented formula vs. a standard formula toward the pursuit of breastfeeding | 3 months of age
Describe the growth, according to the nutrition group | 3 and 5 months of age
Describe the milk tolerance at the weaning according to the nutrition group | 3 and 5 months of age
Describe the infection signs according to the nutrition group | 3 and 5 months of age
Describe weight and height, current alimentation and potential infectious diseases since the visit at 5 months of age, according to the nutrition group | 9 months of age
Compare the effect on enterobacteria, clostridium and bifidobacteria of a fermented formula vs. a standard formula toward the pursuit of breastfeeding | 5 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Kalach, MD, Principal Investigator — Hopital Saint Vincent de Paul
Locations (6):
- France (6):
  - Cabinet médical, Bondues
  - Cabinet médical, Dunkirk
  - Cabinet medical, Lambersart
  - Cabinet médical, Lille
  - Hôpital saint Vincent de Paul, Lille
  - Cabinet médical, Roncq